CLINICAL TRIAL: NCT01065311
Title: Mindfulness-based Cognitive Therapy for Chronic Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Michalak (Other)
Responsible Party: Sponsor-Investigator, Johannes Michalak, Prof. Dr. phil., Ruhr University of Bochum
Organization: Ruhr University of Bochum (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFG Mi 700/4
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Major Depression
Keywords: Depressive Disorder; Psychotherapy
MeSH Terms: conditions — Depressive Disorder | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness-based Cognitive Therapy (Experimental): Mindfulness-based Cognitive Therapy is based on an integration of certain aspects of cognitive behavioral therapy for depression (Beck et al., 1979) and components of the Mindfulness-based Stress Reduction program developed by Kabat-Zinn and colleagues (Kabat-Zinn, 1990). After an initial orientation session, the MBCT program is delivered weekly by an instructor in eight 2.5 hr group sessions.
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy; Biological: Standard psychiatric care
- CBASP (Active Comparator): The Cognitive Behavioral Analysis System of Psychotherapy integrates behavioral, cognitive, and interpersonal strategies. After two initial orientation sessions, the MBCT program is delivered by an instructor in eight weekly 2.5 hr group sessions.
  Interventions: Behavioral: The Cognitive Behavioral Analysis System of Psychotherapy; Biological: Standard psychiatric care
- Treatment-as-usual (Active Comparator): Standard psychiatric outpatient care:
  All patients were requested to get treated individually either by a psychiatrist or by a licensed psychotherapist (not member of the study team). If patients were already in psychiatric/psychotherapeutic individual treatment at study intake they continued their treatment with this psychiatrist/psychotherapist
  Interventions: Biological: Standard psychiatric care

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy — Mindfulness-based Cognitive Therapy is based on an integration of aspects of cognitive behavioral therapy for depression (Beck et al., 1979) with components of the Mindfulness-based Stress Reduction program developed by Kabat-Zinn and colleagues (Kabat-Zinn, 1990). After an initial orientation session, the MBCT program is delivered by an instructor in eight weekly 2.5 hr group sessions
  Arms: Mindfulness-based Cognitive Therapy
Behavioral: The Cognitive Behavioral Analysis System of Psychotherapy — The Cognitive Behavioral Analysis System of Psychotherapy integrates behavioral, cognitive, and interpersonal strategies. After two initial orientation sessions, the MBCT program is delivered weekly by an instructor in eight 2.5 hr group sessions.
  Arms: CBASP
Biological: Standard psychiatric care — Antidepressant medication and medical care.
  Standard psychiatric outpatient care:
  All patients were requested to get treated individually either by a psychiatrist or by a licensed psychotherapist (not member of the study team). If patients were already in psychiatric/psychotherapeutic individual treatment at study intake they continued their treatment with this psychiatrist/psychotherapist
  Other Names: Psychiatric care; neurologic care; ambulant setting

SUMMARY:
The propose of the study is to investigate the efficacy of Mindfulness-based Cognitive Therapy (MBCT, Segal, Williams, & Teasdale, 2002) for patients suffering from Chronic Major Depression. The efficacy of MBCT will be compared with the Cognitive Behavioral Analysis System of Psychotherapy (McCullough, 2003), a treatment approach, which has proven it's efficacy yet, and with a treatment-as-usual condition (standard psychiatric outpatient care).

DETAILED DESCRIPTION:
Cognitive Behavioral Analysis System of Psychotherapy (CBASP) is a treatment approach specifically developed for the treatment of chronic depression. CBASP aims to change dysfunctional interpersonal patterns. Mindfulness-based Cognitive Therapy (MBCT) has recently been proposed as a further treatment option for chronic depression. MBCT trains patients to step out of negative ruminative states of mind. There are no direct comparisons of the psychological treatment options for chronic depression.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnoses of Major Depression, single episode, chronic or
* Major Depression, recurrent, chronic
* Hamilton Rating Scale for Depression score > 14
* Beck Depression Inventory II score > 14

Exclusion Criteria:

* History of Schizophrenia or Schizoaffective Disorder
* Current Substance Dependence or Eating Disorder
* Mental Disorder Due to General Medical Condition
* Borderline Personality Disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | Change from Baseline in HAM-D at 8 weeks

SECONDARY OUTCOMES:
Beck Depression Inventory II | Change from Baseline in BDI-II at 8 weeks
Social Adaption Self-evaluation Scale | Change from Baseline in SASS at 8 weeks
Short Form (36) Health Survey | Change from Baseline in SF-36 at 8 weeks
Global Assessment of Functioning Scale | Change from Baseline in HAM-D at 8 weeks
Response Styles Questionnaire | Change from Baseline in RSQ at 8 weeks
Beck Depression Inventory II | Change from Baseline in BDI-II at 6 months
Social Adaption Self-evaluation Scale | Change from Baseline in SASS at 6 months
Short Form (36) Health Survey | Change from Baseline in SF-36 at 6 months
Global Assessment of Functioning Scale | Change from Baseline in GAF at 6 months
Response Styles Questionnaire | Change from Baseline in RSQ at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Michalak, PD Dr. phil., Principal Investigator — University of Hildesheim
Locations (1):
- University of Hildesheim, Hildesheim, Germany

REFERENCES:
- [Derived] Forkmann T, Brakemeier EL, Teismann T, Schramm E, Michalak J. The Effects of Mindfulness-Based Cognitive Therapy and Cognitive Behavioral Analysis System of Psychotherapy added to Treatment as Usual on suicidal ideation in chronic depression: Results of a randomized-clinical trial. J Affect Disord. 2016 Aug;200:51-7. doi: 10.1016/j.jad.2016.01.047. Epub 2016 Apr 19. PMID 27128357
- [Derived] Michalak J, Schultze M, Heidenreich T, Schramm E. A randomized controlled trial on the efficacy of mindfulness-based cognitive therapy and a group version of cognitive behavioral analysis system of psychotherapy for chronically depressed patients. J Consult Clin Psychol. 2015 Oct;83(5):951-63. doi: 10.1037/ccp0000042. Epub 2015 Aug 10. PMID 26371617